CLINICAL TRIAL: NCT04661033
Title: A Multicenter, Open-label, Non-randomized, Phase 1b/2 Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Subcutaneous Isatuximab in Adults With Warm Autoimmune Hemolytic Anemia
Brief Title: Safety, Pharmacokinetics, and Efficacy of Subcutaneous Isatuximab in Adults With Warm Autoimmune Hemolytic Anemia (wAIHA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinuation based on strategic sponsor decision; not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16832; U1111-1255-5350 (Registry Identifier: ICTRP); 2020-003880-24 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Warm Autoimmune Hemolytic Anemia (wAIHA)
Keywords: (wAIHA)
MeSH Terms: interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 (Experimental): Participants received 2 doses of Isatuximab 140 milligrams (mg) (1 milliliter [mL]) via subcutaneous (SC) injection every 2 weeks (Q2W) on Day 1 and Day 15.
  Interventions: Drug: Isatuximab SAR650984
- Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 (Experimental): Participants received 6 doses of Isatuximab 280 mg (2 mL) via SC injection Q2W through Day 71.
  Interventions: Drug: Isatuximab SAR650984
- Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 (Experimental): Participants received 6 doses of Isatuximab 560 mg (4 mL) via SC injection Q2W through Day 71.
  Interventions: Drug: Isatuximab SAR650984
- Part B: Isatuximab up to 560 mg SC Q2W x6 (Experimental): Participants were planned to receive 6 doses of Isatuximab up to 560 mg (4 mL) via SC injection Q2W through Day 71
  Interventions: Drug: Isatuximab SAR650984

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form:Solution for injection Route of administration: Subcutaneous

SUMMARY:
Primary Objectives:

* Part A: To evaluate the safety and tolerability of subcutaneous injections of isatuximab in adults with wAIHA
* Part B: To evaluate the efficacy of the selected dose in adults with wAIHA

Secondary Objectives:

* Part A (Cohorts 2 and 3 only)
* To evaluate the efficacy of isatuximab in adults with wAIHA
* To evaluate the durability of response to isatuximab and time to response
* To evaluate the impact of isatuximab treatment on fatigue

Part B

* To evaluate the safety and tolerability of isatuximab in adults with wAIHA
* To evaluate the durability of response to isatuximab and time to response
* To evaluate the impact of isatuximab treatment on fatigue

Parts A (all Cohorts) and B

* To evaluate the effect of isatuximab on markers of hemolysis
* To characterize the pharmacokinetic profile of isatuximab in adults with wAIHA
* To evaluate the immunogenicity of isatuximab

DETAILED DESCRIPTION:
28 weeks (including screening)

ELIGIBILITY:
Inclusion criteria :

* Participant must be ≥18 to years of age, inclusive, at the time of signing the informed consent.

  - Males and females with a confirmed diagnosis of primary w AIHA or systemic lupus erythematosus (SLE)-associated w AIHA (without other SLE-related manifestations apart from cutaneous and musculoskeletal manifestations) who meet the following criteria:
  1. Hemoglobin level <10 g/dL at screening.
  2. Hemolysis (haptoglobin ≤40 mg/dL and total or indirect/unconjugated bilirubin above the upper limit of normal).
  3. Positive direct antiglobulin test (DAT) (IgG or IgG + complement C3d pattern or IgM warm autoantibodies (positive dual DAT)).

     * Participants who have previously failed to maintain a sustained response after treatment with corticosteroids (corticosteroid-refractory or corticosteroid-dependent primary wAIHA).
     * Part A only: Participants who have previously failed to maintain a sustained response after treatment with rituximab (or other anti-CD20 monoclonal antibodies). The last dose of the anti-CD20 antibody must have been administered at least 12 weeks before enrollment.
     * Part B: Participants who have had an insufficient response to at least 1 prior therapy in addition to corticosteroids (splenectomy is regarded as a prior therapy).
     * Contraceptive use by men and women

     Exclusion criteria:
* Clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the participant or compromise the quality of the data derived from his or her participation in the study as determined by the Investigator.

  * Serious infection that required hospitalization within 3 months prior to enrollment.
  * Secondary wAIHA from any cause including drugs, lymphoproliferative disorders, infectious or autoimmune disease (SLE without other SLE-related manifestations apart from cutaneous and musculoskeletal manifestations is allowed), or active hematologic malignancies. Participants with positive antinuclear antibodies but without a definitive diagnosis of an autoimmune disease are allowed.
  * History of coagulation or bleeding disorders (Evans Syndrome is allowed).
  * Uncontrolled or active HBV or HCV infection
  * HIV infection.
  * Serum gammaglobulin levels <3 g/L.
  * Females who are pregnant, lactating, or considered unreliable with respect to contraceptive practice.
  * Concurrent treatment with corticosteroids, unless the participant has been on a stable daily dose for ≥ 15 days prior to enrollment.
  * Treatment with cyclophosphamide within 4 weeks prior to enrollment.
  * Treatment with cytotoxic drugs (other than cyclophosphamide) within 12 weeks prior to enrollment.
  * Treatment with non-cytotoxic, immunomodulatory drugs (including but not limited to Cyclosporine, Sirolimus, Tacrolimus, Idelalisib, Ibrutinib), excluding biologic agents, within 4 weeks prior to enrollment.
  * Treatment with any biologic agent within 12 weeks prior to enrollment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Fox Chase Cancer Center Site Number : 8400004, Philadelphia, Pennsylvania, United States
- Investigational Site Number : 2500001, Créteil, France
- Investigational Site Number : 2760001, Essen, Germany
- Investigational Site Number : 3800001, Milan, Italy
- Investigational Site Number : 5280001, Leiden, Netherlands
- Investigational Site Number : 8260001, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16832 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25198&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in 6 countries. A total of 10 participants were screened from 09 September 2021 to 19 December 2022, of which 2 participants were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 8 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled in the study and included in 3 Cohorts in Part A. The study was prematurely terminated based on strategic sponsor decision during Part A; not driven by any safety concerns. Hence Part B was not conducted, and no analysis was performed.
Period: Overall Study
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 | Part B: Isatuximab up to 560 mg SC Q2W x6
Started | 3 | 3 | 2 | 0
Participants Who Completed the Study Treatment Period | 3 | 2 | 1 | 0
Completed | 0 | 3 | 1 | 0
Not Completed | 3 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Switch of cohort due to retreatment criteria met | 1 | 0 | 0 | 0
Not completed — As per Principal Investigator (PI) decision | 1 | 0 | 0 | 0
Not completed — Early discontinuation as per PI | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants exposed to the investigational medicinal product (IMP) (regardless of the amount of treatment administered). The study was prematurely terminated based on strategic sponsor decision during Part A; not driven by any safety concerns, hence Part B was not conducted, and no analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 | Part B: Isatuximab up to 560 mg SC Q2W x6 | Total
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (24.7) | 44.7 (7.6) | 47.5 (30.4) |  | 50.9 (19.3)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 1 | 3 | 1 | 0 | 5
  65 to 84 years | 2 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 5
  Male | 2 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 2 | 0 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) And Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is defined as an AE that occurred from the time of the first IMP administration up to 30 days (included) after the last IMP administration. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From first dose of study drug (Day 1) up to 30 days after last study intervention administration, approximately 101 days
Population: Safety Population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants
  Any TEAEs | 2 | 2 | 2
  Any TESAEs | 1 | 0 | 1

2. Primary Outcome: Part A: Number of Participants With Potentially Clinically Significant Abnormality (PCSA): Hematology
Description: Blood samples were collected to determine the hematology laboratory significant abnormalities. PCSA values: abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Hemoglobin (Hb): ≤ 115 grams per Liter (g/L) (Male[M]); ≤ 95 g/L (Female[F]), ≥ 185 g/L (M); ≥ 165 g/L (F), Decrease from baseline ≥ 20 g/L; Hematocrit: ≤ 0.37 volume per volume (v/v) (M); ≤ 0.32 v/v (F), ≥ 0.55 v/v (M); ≥ 0.5 v/v (F); Erythrocyte Count: ≥ 6 x 10^12 per Liter (/L); Platelet count: < 100 x 10^9/L, ≥ 700 x 10^9/L; Leukocytes: < 3 x 10^9/L (Non-Black [NB]); < 2 x 10^9/L (Black [B]), ≥ 16 x 10^9/L; Neutrophils: < 1.5 x 10^9/L (B); < 1 x 10^9/L (B); Lymphocytes: > 4 x 10^9/L; Monocytes: > 0.7 x 10^9/L; Basophils: > 0.1 x 10^9/L; Eosinophils: > 0.5 x 10^9/L or > Upper limit of Normal (ULN) (if ULN ≥ 0.5 x 10^9/L).
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: Safety Population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants
  Hb: ≤ 115 g/L (M); ≤ 95 g/L (F) | 3 | 3 | 2
  Hb: ≥ 185 g/L (M); ≥ 165 g/L (F), | 0 | 0 | 0
  Hb: Decrease from baseline ≥ 20 g/L | 0 | 1 | 0
  Hematocrit: ≤ 0.37 v/v (M); ≤ 0.32 v/v (F) | 3 | 3 | 2
  Hematocrit: ≥ 0.55 v/v (M); ≥ 0.5 v/v (F) | 0 | 0 | 0
  Erythrocyte Count: ≥ 6 x 10^12/L | 0 | 0 | 0
  Platelet Count: < 100 x 10^9/L | 0 | 0 | 0
  Platelet Count: ≥ 700 x 10^9/L | 0 | 1 | 0
  Leukocytes: < 3 x 10^9/L (NB); < 2 x 10^9/L (B) | 0 | 0 | 1
  Leukocytes: ≥ 16 x 10^9/L | 2 | 1 | 1
  Neutrophils: < 1.5 x 10^9/L (NB); < 1 x 10^9/L (B) | 0 | 0 | 1
  Lymphocytes: > 4 x 10^9/L | 1 | 0 | 0
  Monocytes: > 0.7 x 10^9/L | 2 | 1 | 1
  Basophils: > 0.1 x 10^9/L | 2 | 1 | 1
  Eosinophils: > 0.5 x 10^9/L or > ULN (if ULN ≥ 0.5 x 10^9/L) | 1 | 0 | 1

3. Primary Outcome: Part A: Number of Participants With PCSA: Clinical Chemistry And Electrolyte Parameters
Description: Blood samples were collected to determine the clinical chemistry laboratory and electrolyte parameters significant abnormalities. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Glucose: ≤ 3.9 millimoles per Liter (mmol/L) and < Lower limit of normal (LLN), ≥ 11.1 mmol/L (unfasted); ≥ 7 mmol/L (fasted); Creatinine: ≥ 150 micromoles (µmol)/L, ≥ 30% change from baseline, ≥ 100% change from baseline, Alanine Aminotransferase (ALT): > 3 ULN, > 5 ULN, > 10 ULN; Aspartate Aminotransferase (AST): > 3 ULN; Alkaline Phosphatase (ALP): > 1.5 ULN; Total Bilirubin: > 1.5 ULN, > 2 ULN; Sodium: ≤ 129 mmol/L, ≥ 160 mmol/L and Potassium: < 3 mmol/L, ≥ 5.5 mmol/L.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: Safety Population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants
  Glucose: ≤ 3.9 mmol/L and < LLN | 0 | 0 | 1
  Glucose: ≥ 11.1 mmol/L (unfasted); ≥ 7 mmol/L (fasted) | 0 | 1 | 0
  Creatinine: ≥ 150 µmol/L | 0 | 0 | 0
  Creatinine: ≥ 30% change from baseline | 2 | 0 | 0
  Creatinine: ≥ 100% change from baseline | 1 | 0 | 0
  ALT: > 3 ULN | 1 | 0 | 1
  ALT: > 5 ULN | 1 | 0 | 0
  ALT: > 10 ULN | 0 | 0 | 0
  AST: > 3 ULN | 0 | 0 | 0
  ALP: > 1.5 ULN | 0 | 0 | 0
  Total Bilirubin: > 1.5 ULN | 3 | 2 | 2
  Total Bilirubin: > 2 ULN | 3 | 2 | 2
  Sodium: ≤ 129 mmol/L | 0 | 0 | 0
  Sodium: ≥ 160 mmol/L | 0 | 0 | 0
  Potassium: < 3 mmol/L | 0 | 0 | 0
  Potassium: ≥ 5.5 mmol/L | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Potentially Clinically Significant Abnormality: Urinalysis
Description: Urine samples were collected to determine the urinalysis parameter significant abnormalities. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: pH: ≤ 4.6 or ≥ 8.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: Safety Population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants
  pH: ≤ 4.6 | 0 | 0 | 0
  pH: ≥ 8 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Potentially Clinically Significant Abnormality: Vital Signs
Description: Vital signs were examined to determine the abnormalities. Vital signs included Sitting systolic blood pressure (SSBP), Sitting diastolic blood pressure (SDBP), Sitting heart rate (SHR) and weight. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: SSBP: ≤95 millimeters of mercury (mmHg) and decrease from baseline ≥20 mmHg; ≥160 mmHg and increase from baseline ≥20 mmHg; SDBP: ≤45 mmHg and decrease from baseline ≥10 mmHg, ≥ 110 mmHg and increase from baseline ≥ 10 mmHg; SHR: ≤ 50 beats per minute (bpm) and decrease from baseline ≥ 20 bpm, ≥120 bpm and increase from baseline ≥ 20 bpm; Weight: ≥ 5% decrease from baseline, ≥5% increase from baseline.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: Safety Population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants
  SSBP: ≤95 mmHg and decrease from baseline ≥20 mmHg | 0 | 0 | 2
  SSBP: ≥160 mmHg and increase from baseline ≥20 mmHg | 1 | 0 | 0
  SDBP: ≤45 mmHg and decrease from baseline ≥10 mmHg | 0 | 0 | 2
  SDBP: ≥ 110 mmHg and increase from baseline ≥ 10 mmHg | 0 | 0 | 0
  SHR: ≤ 50 bpm and decrease from baseline ≥ 20 bpm | 0 | 0 | 0
  SHR: ≥ 120 bpm and increase from baseline ≥ 20 bpm | 0 | 0 | 1
  Weight: ≥5% decrease from baseline | 0 | 0 | 0
  Weight: ≥ 5% increase from baseline | 1 | 0 | 1

6. Primary Outcome: Part B: Overall Response Rate (Response [R] Or Complete Response [CR]) At Day 85
Description: Overall response rate was defined as the percentage of participants with a response (R) or complete response (CR) over the evaluable participants. R was defined as an increase in Hb by ≥2 g/dL from baseline and an absence of transfusion in the last 7 days and absence of rescue medications in the past 4 weeks. Biochemical evidence of hemolysis might still be present. CR was defined as Hb ≥11 g/dL (women) or ≥12 g/dL (men), no evidence of hemolysis (normal bilirubin, Lactate dehydrogenase [LDH], haptoglobin, and reticulocytes), and absence of transfusion in the last 7 days and absence of rescue medication in the past 4 weeks.
Time Frame: Day 85
Population: The study was prematurely terminated based on strategic sponsor decision during Part A; not driven by any safety concerns, hence Part B was not conducted, and no analysis was performed.
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

7. Secondary Outcome: Part A: Cohorts 2 and 3: Overall Response Rate (Response [R] Or Complete Response [CR]) At Day 85 And Day 169
Description: Overall response rate was defined as the percentage of participants with a R or CR over the evaluable participants. R was defined as an increase in Hb by ≥2 g/dL from baseline and an absence of transfusion in the last 7 days and absence of rescue medications in the past 4 weeks. Biochemical evidence of hemolysis might still be present. CR was defined as Hb ≥11 g/dL (women) or ≥12 g/dL (men), no evidence of hemolysis (normal bilirubin, LDH, haptoglobin, and reticulocytes), and absence of transfusion in the last 7 days and absence of rescue medication in the past 4 weeks
Time Frame: Day 85 and Day 169
Population: Efficacy population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 2
Percentage of participants
  Day 85 | 0.0 | 50.0
  Day 169 | 0.0 | 0.0

8. Secondary Outcome: Part A: Cohorts 2 and 3: Percentage Of Participants With Durable Hemoglobin (Hb) Response By Day 169
Description: Durable response was defined as Hb level ≥10 g/dL with an increase from baseline of ≥2 g/dL on three consecutive evaluable visits during the study period; with absence of transfusion and no rescue medication during the period of 3 consecutive visits and for at least 7 days (transfusions) and 4 weeks (rescue medication) prior to the first consecutive visit.
Time Frame: From first dose of study drug (Day 1) up to end of study (Day 169)
Population: Efficacy population included all participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 2
Percentage of participants | 0 | 50

9. Secondary Outcome: Part A: Cohorts 2 and 3: Absolute Change From Baseline in Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Scale Score At Day 85 and Day 169
Description: The FACIT-Fatigue scale is a 13-item questionnaire assessing fatigue where participants scored each item on a 5-point scale (0 to 4): 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52, where higher score (and positive change scores) indicated better functioning. Baseline was defined as the Day 1 pre-dose value.
Time Frame: Baseline (Day 1), Day 85 and Day 169
Population: Efficacy population included all participants exposed to the IMP (regardless of the amount of treatment administered). Only those participants with data collected at each specified timepoint are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 2
Score on a scale
  Day 85: number analyzed (Participants) | 3 | 1
  Day 85 | 7.3 (9.3) | 12.0 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Day 169: number analyzed (Participants) | 1 | 1
  Day 169 | 1.0 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | 4.0 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

10. Secondary Outcome: Part A: Absolute Change From Baseline In Lactate Dehydrogenase (LDH) at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were collected to evaluate the effect of Isatuximab on marker of hemolysis: LDH. Baseline is defined as the last assessment value before IMP.
Time Frame: Cohort 1 : Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, and 12; Cohorts 2 and 3: Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
International Units per Liter (IU/L)
  Pre-dose at Week 1 | 84.0 (347.5) | -67.3 (81.4) | -264.0 (196.6)
  Pre-dose at Week 2: number analyzed (Participants) | 2 | 3 | 2
  Pre-dose at Week 2 | 13.0 (192.3) | -110.7 (126.5) | -331.5 (236.9)
  Pre-dose at Week 4 | -342.3 (130.2) | -124.0 (133.3) | -234.5 (105.4)
  Pre-dose at Week 8: number analyzed (Participants) | 2 | 3 | 2
  Pre-dose at Week 8 | -355.5 (444.8) | -136.0 (349.9) | -309.5 (231.2)
  Pre-dose at Week 12: number analyzed (Participants) | 2 | 3 | 1
  Pre-dose at Week 12 | -134.0 (183.8) | -22.0 (201.8) | -146.0 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 24: number analyzed (Participants) | 0 | 3 | 1
  Pre-dose at Week 24 |  | 278.7 (601.0) | -135.0 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

11. Secondary Outcome: Part A: Absolute Change From Baseline In Haptoglobin at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were collected to evaluate the effect of Isatuximab on marker of hemolysis: Haptoglobin. Baseline was defined as the last assessment value before IMP.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Grams per Liter (g/L)
  Pre-dose at Week 1 | 0.000 (0.000) | 0.030 (0.026) | -0.005 (0.007)
  Pre-dose at Week 2: number analyzed (Participants) | 2 | 3 | 1
  Pre-dose at Week 2 | 0.000 (0.000) | 0.000 (0.000) | -0.010 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 4: number analyzed (Participants) | 2 | 3 | 2
  Pre-dose at Week 4 | 0.000 (0.000) | -0.016 (0.028) | -0.005 (0.007)
  Pre-dose at Week 8: number analyzed (Participants) | 2 | 2 | 2
  Pre-dose at Week 8 | 0.000 (0.000) | -0.025 (0.035) | 2.995 (4.250)
  Pre-dose at Week 12: number analyzed (Participants) | 1 | 2 | 1
  Pre-dose at Week 12 | 0.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -0.025 (0.035) | -0.010 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 24: number analyzed (Participants) | 0 | 2 | 1
  Pre-dose at Week 24 |  | -0.022 (0.038) | -0.050 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

12. Secondary Outcome: Part A: Absolute Change From Baseline In Reticulocytes at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were collected to evaluate the effect of Isatuximab on marker of hemolysis: Reticulocytes. Baseline was defined as the last assessment value before IMP.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 1 | 3 | 1
10^9 cells per Liter
  Pre-dose at Week 1 | 86.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -25.533 (49.878) | -158.400 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 2 | 43.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -29.733 (36.258) | -347.400 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 4 | -51.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -36.833 (34.662) | -370.300 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 8 | -9.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -31.733 (84.835) | -280.300 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 12 | 44.000 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | -6.133 (33.198) | -250.600 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 24: number analyzed (Participants) | 0 | 3 | 1
  Pre-dose at Week 24 |  | -126.933 (70.273) | 9.900 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

13. Secondary Outcome: Part A: Absolute Change From Baseline In Total Bilirubin at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were collected to evaluate the effect of Isatuximab on marker of hemolysis: Total Bilirubin. Baseline was defined as the last assessment value before IMP.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (μmol/L)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Micromoles per Liter (μmol/L)
  Pre-dose at Week 1 | -8.52 (19.00) | -7.01 (3.12) | -15.00 (2.83)
  Pre-dose at Week 2 | 2.45 (15.88) | -6.38 (1.10) | -13.00 (4.24)
  Pre-dose at Week 4 | -18.26 (31.86) | -2.00 (1.78) | -8.50 (7.78)
  Pre-dose at Week 8 | -14.31 (5.89) | -8.21 (17.53) | -14.50 (10.61)
  Pre-dose at Week 12: number analyzed (Participants) | 3 | 3 | 1
  Pre-dose at Week 12 | 0.70 (18.47) | 3.65 (11.83) | -4.00 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.
  Pre-dose at Week 24: number analyzed (Participants) | 0 | 3 | 1
  Pre-dose at Week 24 |  | 0.06 (9.08) | 17.00 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

14. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) Of Isatuximab
Description: Blood samples were collected at the specified timepoints. Cmax was defined as maximum concentration observed after the first infusion. The non-compartmental pharmacokinetic (PK) analysis was performed.
Time Frame: Post-dose on Day 1
Population: Pharmacokinetic (PK) population included all participants exposed to the IMP (regardless of the amount of treatment administered), without any major or critical deviations related to IMP administration and for whom the PK data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Micrograms per milliliter (μg/mL) | 3.64 (1.19) | 7.41 (6.29) | 151 (121)

15. Secondary Outcome: Part A: Time to Reach Cmax (Tmax) of Isatuximab
Description: Blood samples were collected at the specified timepoints. Tmax was defined as time to reach Cmax. The non-compartmental PK analysis was performed.
Time Frame: Post-dose on Day 1
Population: PK population included all participants exposed to the IMP (regardless of the amount of treatment administered), without any major or critical deviations related to IMP administration and for whom the PK data were considered sufficient and interpretable.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Hours (h) | 89.50 [89.35 to 96.33] | 92.68 [48.58 to 119.17] | 202.69 [94.80 to 310.58]

16. Secondary Outcome: Part A: Area Under the Plasma Concentration Versus Time Curve Calculated Using the Trapezoidal Method From Time Zero to Time of the Last Concentration Observed Above the Lower Limit of Quantification (Clast) (AUClast) of Isatuximab
Description: Blood samples were collected at the specified timepoints. AUClast was defined as area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to time of the Clast. The non-compartmental PK analysis was performed.
Time Frame: Post-dose on Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter(h*μg/mL)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Hours*micrograms per milliliter(h*μg/mL) | 540 (30.0) | 879 (99.0) | 23900 (41.0)

17. Secondary Outcome: Part A: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval (AUCtau) of Isatuximab
Description: Blood samples were collected at the specified timepoints. AUCtau was defined as area under the plasma concentration versus time curve over the dosing interval. The non-compartmental PK analysis was performed.
Time Frame: Post-dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter(h*μg/mL)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 1
Hours*micrograms per milliliter(h*μg/mL) | 560 (171) | 1370 (1350) | 17800 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

18. Secondary Outcome: Part A: Mean Plasma Trough Concentration Of Isatuximab
Description: Blood samples were collected at the specified timepoints. The non-compartmental Pharmacokinetic (PK) analysis was performed
Time Frame: Post-dose on Days 15, 29, 43 and 57
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Micrograms per milliliter (μg/mL)
  Day 15 | 0.0114 (0.0140) | 0.678 (0.994) | 140 (137)
  Day 29 | 0.167 (0.270) | 7.30 (7.13) | 134 (62.3)
  Day 43 | 0.00111 (0.00131) | 6.69 (5.90) | 62.0 (87.7)
  Day 57: number analyzed (Participants) | 3 | 2 | 1
  Day 57 | NA (NA) — Mean and Standard deviation could not be determined as the values were below the lower limit of quantification (LLOQ). LLOQ was 0.0005 µg/mL | 10.7 (4.08) | 146 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

19. Secondary Outcome: Part A: Number Of Participants With Anti-Isatuximab Antibodies
Description: Plasma samples were collected to evaluate antibodies to Isatuximab. Plasma samples were screened for antibodies binding to Isatuximab. Post-baseline positive, defined as Anti-drug antibody (ADA) that developed at any time during the ADA on-study observation period in participants without pre-existing ADA. Number of participants with positive ADA have been reported.
Time Frame: Up to Days 169
Population: ADA population included all participants exposed to the IMP (regardless of the amount of treatment administered) with at least one evaluable ADA sample (positive, negative or inconclusive) during the treatment emergent (TE) period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6
Number analyzed (Participants) | 3 | 3 | 2
Participants | 1 | 1 | 0

20. Secondary Outcome: Part B: Number of Participants With TEAEs And TESAEs
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is defined as an AE that occurred from the time of the first IMP administration up to 30 days (included) after the last IMP administration. A SAE is defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

21. Secondary Outcome: Part B: Number of Participants With PCSA: Hematology
Description: Blood samples were planned to be collected to determine the hematology laboratory significant abnormalities. PCSA values: abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Hb: ≤ 115 g/L (M); ≤ 95 g/L (F), ≥ 185 g/L (M); ≥ 165 g/L (F), Decrease from baseline ≥ 20 g/L; Hematocrit: ≤ 0.37 v/v (M); ≤ 0.32 v/v (F), ≥ 0.55 v/v (M); ≥ 0.5 v/v (F); Erythrocyte Count: ≥ 6 x 10^12/L); Platelet count: < 100 x 10^9/L, ≥ 700 x 10^9/L; Leukocytes: < 3 x 10^9/L (NB); < 2 x 10^9/L (B), ≥ 16 x 10^9/L; Neutrophils: < 1.5 x 10^9/L (B); < 1 x 10^9/L (B); Lymphocytes: > 4 x 10^9/L; Monocytes: > 0.7 x 10^9/L; Basophils: > 0.1 x 10^9/L; Eosinophils: > 0.5 x 10^9/L or > ULN (if ULN ≥ 0.5 x 10^9/L).
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

22. Secondary Outcome: Part B: Number of Participants With PCSA: Clinical Chemistry And Electrolyte Parameters
Description: Blood samples were planned to be collected to determine the clinical chemistry laboratory and electrolyte parameters significant abnormalities. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Glucose: ≤ 3.9 mmol/L and < LLN, ≥ 11.1 mmol/L (unfasted); ≥ 7 mmol/L (fasted); Creatinine: ≥ 150 µmol/L, ≥ 30% change from baseline, ≥ 100% change from baseline, ALT: > 3 ULN, > 5 ULN, > 10 ULN; AST: > 3 ULN; ALP: > 1.5 ULN; Total Bilirubin: > 1.5 ULN, > 2 ULN; Sodium: ≤ 129 mmol/L; ≥ 160 mmol/L; Potassium: < 3 mmol/L, ≥ 5.5 mmol/L and Calcium
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

23. Secondary Outcome: Part B: Number of Participants With Potentially Clinically Significant Abnormality: Urinalysis
Description: Urine samples were planned to be collected to determine the urinalysis parameter significant abnormalities. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: pH ≤ 4.6 or ≥ 8.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

24. Secondary Outcome: Part B: Number of Participants With Potentially Clinically Significant Abnormality: Vital Signs
Description: Vital signs were planned to be examined to determine the abnormalities. Vital signs included SSBP, SDBP, SHR and weight. PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: SSBP: ≤ 95 mmHg and decrease from baseline ≥ 20 mmHg, ≥ 160 mmHg and increase from baseline ≥20 mmHg; SDBP: ≤ 45 mmHg and decrease from baseline ≥ 10 mmHg, ≥ 110 mmHg and increase from baseline ≥ 10 mmHg; SHR: ≤ 50 bpm and decrease from baseline ≥ 20 bpm, ≥ 120 bpm and increase from baseline ≥ 20 bpm; Weight: ≥ 5% decrease from baseline, ≥5% increase from baseline.
Time Frame: From first dose of study drug (Day 1) up to end of study, approximately 169 days
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

25. Secondary Outcome: Part B: Percentage Of Participants With Durable Hemoglobin Response By Day 169
Description: as for outcome 8
Time Frame: From first dose of study drug (Day 1) up to end of study (Day 169)
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

26. Secondary Outcome: Part B: Overall Response Rate (Response [R] Or Complete Response [CR]) At Day 169
Description: as for outcome 7
Time Frame: Day 169
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

27. Secondary Outcome: Part B: Absolute Change From Baseline In FACIT-Fatigue Scale Score At Day 85 And Day 169
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Day 85 and Day 169
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

28. Secondary Outcome: Part B: Absolute Change From Baseline In LDH at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were planned to be collected to evaluate the effect of Isatuximab on marker of hemolysis: LDH. Baseline was defined as the last assessment value before IMP
Time Frame: Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

29. Secondary Outcome: Part B: Absolute Change From Baseline In Haptoglobin at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were planned to be collected to evaluate the effect of Isatuximab on marker of hemolysis: Haptoglobin. Baseline was defined as the last assessment value before IMP
Time Frame: Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

30. Secondary Outcome: Part B: Absolute Change From Baseline In Reticulocytes at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were planned to be collected to evaluate the effect of Isatuximab on marker of hemolysis: Reticulocytes. Baseline was defined as the last assessment value before IMP
Time Frame: Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

31. Secondary Outcome: Part B: Absolute Change From Baseline In Total Bilirubin at 1, 2, 4, 8, 12, and 24 Weeks
Description: Blood samples were planned to be collected to evaluate the effect of Isatuximab on marker of hemolysis: Total Bilirubin. Baseline was defined as the last assessment value before IMP
Time Frame: Baseline (Day 1) and pre-dose at Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

32. Secondary Outcome: Part B: Cmax Of Isatuximab
Description: Blood samples were planned to be collected at the specified timepoints. Cmax was defined as maximum concentration observed after the first infusion.
Time Frame: Post-dose on Day 1
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

33. Secondary Outcome: Part B: AUCtau of Isatuximab
Description: Blood samples were planned to be collected at the specified timepoints. AUCtau was defined as area under the plasma concentration versus time curve over the dosing interval.
Time Frame: Post-dose on Day 1
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

34. Secondary Outcome: Part B: Mean Plasma Trough Concentration Of Isatuximab
Description: Blood samples were planned to be collected at the specified timepoints.
Time Frame: Post-dose on Days 15, 29, 43 and 57
Population: as for outcome 6
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

35. Secondary Outcome: Part B: Number Of Participants With Anti-Isatuximab Antibodies
Description: Plasma samples were planned to be collected to evaluate antibodies to Isatuximab. Plasma samples were planned to be screened for antibodies binding to Isatuximab. Post-baseline positive, defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA.
Time Frame: Up to Days 169
Population: as for outcome 6
Groups:
- Part B: Isatuximab up to 560 mg SC Q2W x6: Participants were planned to receive 6 doses of Isatuximab up to 560 mg (4 mL) via SCinjection Q2W through Day 71.
Arm/Group | Part B: Isatuximab up to 560 mg SC Q2W x6
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first dose of study drug (Day 1) up to 30 days after last study intervention administration, approximately 101 days. All-cause mortality (deaths) were collected from first dose of study drug (Day 1) up to end of study, approximately 169 days.
Description: Analysis was performed on safety population. The study was prematurely terminated based on strategic sponsor decision during Part A; not driven by any safety concerns, hence Part B was not conducted, and no analysis was performed.
Arm/Group | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 | Part B: Isatuximab up to 560 mg SC Q2W x6
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 (N=3) | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 (N=3) | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 (N=2) | Part B: Isatuximab up to 560 mg SC Q2W x6 (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: Isatuximab 140 mg SC Q2W x2 (N=3) | Part A: Cohort 2: Isatuximab 280 mg SC Q2W x6 (N=3) | Part A: Cohort 3: Isatuximab 560 mg SC Q2W x6 (N=2) | Part B: Isatuximab up to 560 mg SC Q2W x6 (N=0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated based on strategic sponsor decision during Part A; not driven by any safety concerns, hence Part B was not conducted, and no analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04661033/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT04661033/SAP_001.pdf